CLINICAL TRIAL: NCT01358058
Title: Phase II Study of Proton Radiation Therapy for Low Grade and Favorable Grade 3 Gliomas
Brief Title: Proton Radiation Therapy for Gliomas
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Helen A. Shih, MD, Attending Radiation Oncologist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-439
Record Dates: First submitted 2011-05-17; First posted 2011-05-23 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Low Grade Glioma; WHO Grade 3 Glioma With IDH1 Mutation; WHO Grade 3 Glioma With 1p/19q Codeletion
Keywords: Brain tumors; Radiation; Proton; Gliomas
MeSH Terms: conditions — Brain Neoplasms; Glioma | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton radiation therapy (Experimental): Single arm study delivering fractionated proton therapy over 6 week (54-59.4 Gy(RBE))
  Interventions: Radiation: Proton radiation

INTERVENTIONS:
Radiation: Proton radiation — Total dose of 54-59.4 Gy(RBE) at 1.8 Gy(RBE) per daily fraction delivered 5 days per week on weekdays for 6-6.5 weeks.

SUMMARY:
In this research study the investigators are looking at a type of radiation called proton radiation. Proton radiation has been shown to deliver virtually no radiation beyond the area of the tumor, sparing surrounding normal tissue from exposure. This may reduce side effects that patients would normally experience with conventional radiation therapy.

In this research study the investigators are looking to determine if proton radiation with a reduced field size will be as effective in controlling tumor growth as photon therapy, while reducing the treatment-related side effects observed in patients with brain tumors.

DETAILED DESCRIPTION:
Proton radiation will be delivered daily for approximately 6 weeks. Subjects will be assessed weekly for side effects. Each visit will take about 15 minutes.

Subjects will have follow-up visits at 3, 6, 12, 24, 36, 48, 60, 72, and 84 months after their last proton radiation treatment. They will receive a physical exam, MRI, have blood tests (about 4 teaspoons) and answer questionnaires regarding medical history, quality of life, and emotional well-being. Subjects will also receive a neurocognitive exam annually.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed low-grade gliomas OR Grade III anaplastic glioma with either or both IDH1 mutation or 1p/19q codeletion
* Subject must be indicated for radiation therapy
* Life expectancy greater than 5 years
* Willing to participate in rigorous neurocognitive evaluations at baseline and serially following treatment
* Able to speak and comprehend English
* Recovered from adverse events due to agents administered more than 4 weeks before entering study
* Able to undergo MRI scans

Exclusion Criteria:

* Prior cranial radiation therapy
* Chemotherapy within 4 weeks prior to entering study
* Pregnant or breastfeeding
* Known brain metastases
* Baseline neurocognitive or emotional disorders
* Uncontrolled intercurrent illness
* History of a different malignancy unless disease-free for at least 5 years
* HIV positive on antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2011-05; Primary Completion 2027-05 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 7 years
  To assess progression free survival of this treatment program.

SECONDARY OUTCOMES:
Safety and Tolerability | 7 years
  To assess the number of participants with late effects from radiation therapy
Overall survival | 7 years
  To assess overall survival of this treatment program.

CONTACTS AND LOCATIONS:
Overall Officials: Helen A Shih, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States